CLINICAL TRIAL: NCT03401476
Title: Effect of Morphine on Dyspnea and 6-Minute Walk Distance in Pulmonary Arterial Hypertension
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: John Granton (Other)
Responsible Party: Sponsor-Investigator, John Granton, Principal Investigator, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MorPHine
Record Dates: First submitted 2017-04-30; First posted 2018-01-17 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morphine sulfate - Visit 1 (Active Comparator): Patients who are randomized to this group will be administered a fixed 5mg dose of oral morphine sulfate prior to performing their 6MWT at Visit 1.
  Interventions: Drug: Morphine Sulfate
- Morphine sulfate - Visit 2 (Active Comparator): Patients who are randomized to this group will be administered a fixed 5mg dose of oral morphine sulfate prior to performing their 6MWT at Visit 2.
  Interventions: Drug: Morphine Sulfate

INTERVENTIONS:
Drug: Morphine Sulfate — Morphine Sulfate Tablets
  Other Names: Statex

SUMMARY:
Despite advances in treatment and corresponding improvements in survival, patients with pulmonary arterial hypertension (PAH) remain highly symptomatic. In one survey of 315 patients with PAH, sixty-eight percent had moderate or severe dyspnea on exertion and 40% had a profound and clinically significant deficit in quality of life. Palliative care is being increasingly investigated in life-limiting cardiovascular diseases to alleviate symptoms. In PAH, its implementation is frequently delayed until end-of-life. Opioids are a common palliative care intervention, however the efficacy and safety of opioids for symptom relief in PAH has not been evaluated.

DETAILED DESCRIPTION:
There is biologic plausibility for opioids in the treatment of dyspnea in PAH. Opioids have widespread effects including venodilation, vasodilation, reducing sympathetic outflow, blunting hypercapnic and hypoxic ventilatory responses, and altering the central perception of dyspnea. Although the origins of dyspnea in PAH are incompletely understood and multifactorial, right ventricular dysfunction reduces exercise capacity and likely also plays a role in the development of dyspnea. Mechanoreceptors situated in the right atrium and right ventricle sense elevated pressures and via sympathetic afferents may lead to an augmentation of ventilatory response and hence dyspnea. Morphine may specifically antagonize this feedback loop by causing venodilation and blunting sympathetics. Morphine also reduces central chemosensitivity and perceptions of dyspnea. Therefore, the drug may antagonize both peripheral and central drivers of dyspnea in PAH.

Investigators will conduct a single-center feasibility study of morphine for treatment of dyspnea and exercise intolerance in PAH. Participants will complete two 6-minute walk tests (6MWT) within one week. Participants will be randomly assigned to receive morphine prior to either the first or second 6MWT. Symptoms and 6-minute walk distance (6MWD) will be compared between the two tests.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* Diagnosis of Group 1 pulmonary hypertension including idiopathic PAH, heritable PAH, and PAH that is drug- or toxin-induced, associated with connective tissue disease, human immunodeficiency virus (HIV) infection, congenital heart disease, or schistosomiasis23
* PAH confirmed by means of a right heart catheterization demonstrating:24

  * Mean pulmonary arterial pressure of ≥ 25 mmHg
  * Pulmonary capillary wedge pressure ≤ 15 mmHg
  * Pulmonary vascular resistance of ≥ 3 Wood units
* World Health Organization (WHO) Functional Class III or ambulatory Class IV
* Six-minute walk test performed within the past 6 months demonstrating a distance of at least 50 metres.
* Unchanged PAH medication regimen for 30 days prior to enrolment. Therapy may include endothelin-receptor antagonists, phosphodiesterase type 5 inhibitors, soluble guanylate cyclase stimulators, or oral or parenteral prostacyclin analogues. Diuretic doses may change.

Exclusion Criteria:

* Group 1 pulmonary hypertension due to portal hypertension
* Group 1 pulmonary hypertension due to pulmonary veno-occlusive disease or pulmonary capillary hemangiomatosis
* Groups 2, 3, 4, or 5 pulmonary hypertension
* Severe renal impairment (estimated glomerular filtration rate < 30 mL/minute/1.73m2 measured within 6 months)
* Severe hepatic impairment (INR > 2.0 in absence of vitamin K antagonist therapy, serum bilirubin > 50mmol/L, cirrhosis on imaging or liver biopsy, prior hepatic encephalopathy, or Model for End-Stage Liver Disease (MELD) score > 19, measured within 6 months, as required based on clinical suspicion)
* Women who are pregnant or breastfeeding (beta-human chorionic gonadotropin (hCG) to confirm non-pregnant status in all females below age 50)
* Hypersensitivity to opioid analgesic, concomitant use with Monoamine Oxidase (MAO) inhibitor or within 14 days of such treatment, concomitant use with barbiturates. Concomitant use with benzodiazepines and/or antipsychotics is permissible provided doses are stable over preceding 1 month.
* Daily use of an opioid-containing medication
* Unstable condition that is a contraindication to opioid use: Central Nervous System (CNS) depression, acute respiratory disease or impairment (acute hypoxia or hypercapnia), acute asthma or Chronic Obstructive Pulmonary Disease (COPD) exacerbation, untreated symptomatic obstructive sleep apnea, unstable cardiac arrhythmias, suspected hypovolemia, recent seizures (within 1 month), active drug abuse, abdominal disease and/or recent GI surgery (within 1 month), active gallbladder disease/biliary colic, untreated depression/suicidality, recent head injury (within 1 month), pre-existing intracranial lesion or increased intracranial pressure, untreated urinary tract obstruction, untreated hypothyroidism, hypopituitarism or Addison's disease.
* Hypotension (resting systolic blood pressure less than or equal to 80mmHg)
* Active or unstable coronary artery disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-05-08 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Borg Dyspnea Score | The Peak Borg Dyspnea Score will be determined over 6 minutes of observation during the conduct of each 6-minute walk test. The 6-minute walk tests and assessments of the peak Borg Dyspnea Score will be recorded within 1 and 7 days of each other.
  Change in peak Borg dyspnea score (morphine versus control)

SECONDARY OUTCOMES:
Change in 6-Minute Walk Distance | The distance travelled during each 6 minute walk will be determined at completion of the 6-minute walk test. The distance travelled during the 6-minute walk test will be recorded within 1 and 7 days of each other.
  Change in six-minute walk distance (morphine versus control)

CONTACTS AND LOCATIONS:
Overall Officials: John Granton, MD, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No